CLINICAL TRIAL: NCT00004638
Title: Immunologic Aspects of the Pathogenesis of Chronic Sinusitis in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Purpose: Diagnostic
Other Study IDs: NCRR-M01RR00069-0609; M01RR000069 (NIH)
Record Dates: First submitted 2000-02-23; First posted 2000-02-24 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-11

CONDITIONS: Sinusitis
Keywords: chronic sinusitis
MeSH Terms: conditions — Sinusitis

INTERVENTIONS:
Procedure: pathogenesis study

SUMMARY:
Chronic sinusitis is a common pediatric disease; it ranks among the top five infectious diseases of the upper respiratory tract. Its treatment is limited and may be due largely in part to a lack of understanding of its cause. The investigators have preliminary data to support the notion that pediatric chronic sinusitis is a distinct disease, different from acute sinusitis and adult chronic sinusitis. We are proposing to perform pathogenesis studies in children with chronic sinusitis. Specifically, we wish to elucidate the microbiologic features and immunologic factors involved in the formation of this disease. The study plan calls for microbiologic (bacterial, viral, and fungal) and immunologic (inflammatory mediators and leukocyte populations) data to be evaluated through a maxillary sinus washing and mucosal biopsies. Four populations will be studied and they are: 10 children with chronic sinusitis, 5 children with acute sinusitis (positive control), 5 children without sinusitis (negative control) and 5 adults with chronic sinusitis (positive secondary control).

ELIGIBILITY:
Inclusion Criteria:

* chronic sinusitis confirmed by imaging study for greater than 12 weeks subjects have failed medical therapy

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital, Denver, Colorado, United States